CLINICAL TRIAL: NCT02187731
Title: FULIMA - A Prospective Study of Dual Time PET/CT and Diffusion Weighted MRI in Multiple Myeloma
Brief Title: Functional Imaging in Multiple Myeloma -PET/CT and Diffusion Weighted Imaging in Multiple Myeloma
Acronym: FULIMA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Brian Oestergaard, MD, Odense University Hospital
Other Study IDs: S-20120209; 13/24748 (Registry Identifier: Danish Dataprotection Agency)
Record Dates: First submitted 2014-04-23; First posted 2014-07-11 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Functional Imaging; PET/CT; Diffusion Weighted MRI
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The FULIMA study is a two-center study at Odense University Hospital and Vejle Hospital, Denmark. The primary objective is to identify the optimal imaging technique for studies in multiple myeloma with focus on PET/CT and MRI.

By combining early (1 hour) and late (3 hours) 18F-2-fluoro-2-deoxy-D- fluorodeoxyglucose(18F-FDG)-PET/CT scans the investigators expect to see increased uptake of radioactive tracer and thus an improved ability to identify malignant tissue. A second tracer 18F-natrium-fluoride is used to explore early signs of bone remodeling. By using new software (ROVER) for interpreting PET data the investigators expect to obtain a quantitative measurement of total disease burden with less risk of misinterpretation of data.

Diffusion weighted MRI (DWI) is a new MRI technique which, like PET/CT, makes it possible quantitatively to calculate the overall disease activity and to give an early evaluation of response to chemotherapy. The study examines DWI for development and standardization.

To validate imaging findings and to explore the pathogenetic heterogeneity of multiple myeloma, the investigators perform CT guided biopsies from PET/ DWI positive sites. Pathoanatomical and immunohistochemical findings and gene expression data from positive sites are compared to random bone marrow. The question is whether disease heterogeneity may explain the lack of FDG uptake in bone marrow in some patients? To the extent that the FULIMA study produces useful data, the defined and standardized imaging techniques will form the basis of a larger prospective study at national level in Denmark.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 50 years at time of signing informed consent.
2. Subject under suspicion of having treatment demanding multiple myeloma in concordance with Danish cancer package criteria
3. Signed informed consent before performance of any study related procedures.
4. Subject is willing and able to comply with the protocol as judged by the investigator.

Exclusion Criteria:

1. Formerly treated multiple myeloma.
2. Known inflammatory disease, recent biological therapies or chemotherapy for non-malignant disease (less than 3 months prior to screening), clinically relevant active infection.
3. Concurrent or recent radiotherapy or surgery less than two weeks prior to screening
4. Glucocorticoid treatment exceeding 10 mg Prednisolone daily, less than two weeks prior to screening.
5. Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at an unacceptable risk if s/he were to participate in the study, e.g. high levels of liver-enzymes and creatinine.
6. Female subject is pregnant or breast feeding.
7. Serious co-morbidity, and other medical or psychiatric illness likely to interfere with participation in this clinical study.
8. Uncontrolled diabetes at the discretion of the investigator.
9. Known or prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer or in situ prostate cancer for which the subject has been disease free for at least three years.
10. POEMS syndrome (plasma cell dyscrasia with poly-neuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes).
11. Exclusion according to MRI procedure (metal implants, claustrophobia, pace-maker).
12. Exclusion according to biopsy study (thrombocytes < 50x /L, activated partial thromboplastin time(APTT) > 40 sec, and international normalized ratio(INR) > 1.5)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective study with 60 patients referred to Haematological Department under the suspicion of having treatment demanding multiple myeloma. Patients will be included from two centres of Haematology.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Multiple myeloma identified as bone disease, myeloma or plasmacytoma | "baseline"
  A 1st complete set of imaging procedures is completed at time of diagnosis "baseline" (week 1-2) for all patients included in the study. The primary hypothesis that 3-hour FDG-PET / CT finds more malignant lesions than the current gold standard procedure, whole body x-ray(WBXR), together with CT and MRI. Concordance analysis will be done by summarizing comparisons of 3-hours FDG-PET/CT versus the remaining modalities. We measure a 95% Wilson-Score Confidence Interval (CI) to demonstrate that 3hours FDG-PET / CT find more malignant lesions than gold standard. This will be concluded at a significance level of 5% if the lower boundary of the 95% CI is larger than 30%.

SECONDARY OUTCOMES:
Disease heterogeneity | Within 2 weeks after imaging procedures
  CT guided or Ultra Sound guided biopsies from PET/ DWI positive sites. Pathoanatomical and immunohistochemical findings and gene expression data from positive sites are compared to random bone marrow.
Early signs of bone remodeling | "baseline", after induction treatment and after end of treatment
  18F-natrium-fluoride-PET/CT is performed at time of diagnosis (baseline) during week 1-2, after induction treatment and after end of treatment. We test if increased 18F-natrium-fluoride uptake is seen in bone sites where, according to CT and DWI, no abnormal bone remodeling is taking place and we observe the association between FDG-PET and fluoride-PET and markers of bone metabolism. We use descriptive statistics for number of bone sites with increased fluoride uptake, 95% Confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Brian Oestergaard, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Derived] Zadeh MZ, Seraj SM, Ostergaard B, Mimms S, Raynor WY, Aly M, Borja AJ, Arani LS, Gerke O, Werner TJ, Zhuang H, Revheim ME, Abildgaard N, Hoilund-Carlsen PF, Alavi A. Prognostic significance of 18F-sodium fluoride in newly diagnosed multiple myeloma patients. Am J Nucl Med Mol Imaging. 2020 Aug 25;10(4):151-160. eCollection 2020. PMID 32929393